CLINICAL TRIAL: NCT00415909
Title: Phase II "Proof of Concept" Study of TALL-104 (MHC Non-Restricted Cytotoxic T-Cell Line) and Imatinib Mesylate (Gleevec) in Chronic Myelogenous Leukemia in Chronic Phase
Brief Title: TALL-104 and Gleevec in Chronic Myelogenous Leukemia Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Abiogen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0837
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Leukemia; Chronic Myelogenous Leukemia; CML; Imatinib; Gleevec; TALL-104
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TALL-104 + IM (Experimental): TALL-104 cells and imatinib mesylate (IM) therapy
  Interventions: Drug: Imatinib Mesylate (IM); Drug: TALL-104 cells

INTERVENTIONS:
Drug: Imatinib Mesylate (IM) — IM Therapy of (100 mg or 400 mg) tablets by mouth, same dose each day.
  Other Names: Gleevec
Drug: TALL-104 cells — TALL-104 cells will be given intravenously over 1 hour at the dose of 109 cells daily for 4 days, on days 1 to 4 of the cycle, and then again on days 7, 10, 14, 17 and 21 of the cycle. One cycle is equal to 28 days. Patients will receive only one cycle of therapy with TALL-104 cells

SUMMARY:
Objectives:

* To determine the response rate and duration of response with combination of TALL-104 cells and imatinib mesylate (IM) therapy in patients with chronic myelogenous leukemia in chronic phase, that have not achieved, or have lost, adequate response to IM.
* To determine the toxicity of the combination of TALL-104 cells and IM therapy in this patient population.

DETAILED DESCRIPTION:
Imatinib mesylate is designed to block the enzyme that is believed to be responsible for starting the type of leukemia patient has. TALL-104 cells are cells of the immune system that have been obtained from a patient with leukemia and then processed in the laboratory to try to make them able to kill leukemia cells.

If found to be eligible to take part in this study, patient will continue receiving imatinib mesylate by mouth at the same schedule and dose patient had been receiving before entering the study. Patient will receive TALL-104 cells through a needle in their vein over 1 hour on Days 1-4, and then again on Days 7, 10, 14, 17, and 21 of the cycle. The cycle will last 28 days.

Blood (about 1 tablespoon) will be drawn every week for the first 4 weeks, then every 2-4 weeks for 2 months, then every 4-6 weeks until 6 months, and then every 3-6 months for routine tests and to check for any effect on organs.

Patient will have follow-up visits at 1 month, 3 months, 6 months, and at least annually for 2 years, and then at least every 5 years from then on for the rest of your life. Blood (about 1 teaspoon) will be drawn to check the status of the disease. An additional 1 tablespoon will also be collected and stored to be analyzed in case unexpected side effects occur after receiving therapy. If patient experiences certain side effects, more blood may need to be drawn and more tests performed based on the side effects experienced.

Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CML in chronic phase who have failed to achieve or have lost an adequate response to IM. For the purpose of this trial this will be defined as a lack of any cytogenetic response after 6 months of therapy or lack of major cytogenetic response after 12 months of therapy with IM. Patients that have lost their major or complete cytogenetic response will also be eligible. Patients who show a sustained increase in breakpoint cluster region gene (BCR)-Abelson gene (ABL)/ABL [BCR-ABL/ABL] ratio of >/= 1-log confirmed in at least two consecutive Polymerase Chain Reaction (PCR) analyses (at least one month apart from each other) will also be eligible.
2. *continued from above: Patients with stable molecular response defined as 2 consecutive PCR-positive results (no more than 1/2 log improvement) will also be eligible. Patients must be taking stable dose of IM for at least 3 months before study enrollment, and recovered from all toxicities related to IM, to grade 0-1.
3. Patients should be in complete or partial hematological remission, including white blood count (WBC) </=20 x 10(9)/L, and platelets </= 600 x 10(9)/L.
4. Eastern Cooperative Oncology Group (ECOG) scale performance status of 2 or less.
5. Age greater than 18 years of age since disease is extremely rare in younger age groups.
6. Adequate liver (total bilirubin of less than 2 times and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) of less than 2 times upper limits of normal), and renal function (creatinine of less than 2 times upper limit of normal).
7. Signed informed consent form.
8. Negative pregnancy test in women of childbearing age.
9. Negative hepatitis B and C screening blood tests.

Exclusion Criteria:

1. Serious intercurrent medical illnesses or active infections requiring parenteral antibiotics that would interfere with the ability of the patient to carry out the treatment program.
2. Female patients who are pregnant or breast-feeding.
3. Patients taking steroids, or those anticipated to receive steroids during the trial therapy.
4. Prior bone marrow transplant.
5. Known positivity for human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 21, 2006 to June 27, 2008.
Groups:
- TALL-104 + IM: TALL-104 cells and imatinib mesylate (IM) therapy. Imatinib Mesylate (IM): IM Therapy of (100 mg or 400 mg) tablets by mouth, same dose each day.
  T Acute Lymphoblastic Leukemia/Lymphoma (TALL)-104 cells: TALL-104 cells will be given intravenously over 1 hour at the dose of 109 cells daily for 4 days, on days 1 to 4 of the cycle, and then again on days 7, 10, 14, 17 and 21 of the cycle. One cycle is equal to 28 days. Patients will receive only one cycle of therapy with TALL-104 cells
Period: Overall Study
Arm/Group | TALL-104 + IM
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Two participants withdrew from the study, and one died of a second, unrelated malignancy.
Arm/Group | TALL-104 + IM
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 65 [54 to 71]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Major and Complete Cytogenetic Response)
Description: Rate is defined as number of participants with response of Major and Complete cytogenetic response out of total study participants. Response evaluated at one and 3 months from start of therapy, then every 3 months in patients with response, for one year, then every 6-12 months. Responses classified according to suppression of Philadelphia (Ph) chromosome by cytogenetic analysis: a) Complete cytogenetic response - Not Ph positive; b) Major cytogenetic response - Ph positive 1-34% of pretreatment value; c) Minor cytogenetic response - Ph positive 35-65% of pretreatment value; d) Minimal cytogenetic response - Ph positive 65-99% of pretreatment value; e) No cytogenetic response - Ph positive 100% of pretreatment value.
Time Frame: Evaluated at baseline (pretreatment) up to 12 months
Population: All three patients received the planned 9 administrations of TALL-104.
Measure: Number; unit: percentage of participants
Arm/Group | TALL-104 + IM
Number analyzed (Participants) | 3
percentage of participants
  Baseline | 0
  1 Month | 67
  3 Months | 33
  12 Months | 33

ADVERSE EVENTS:
Time Frame: Treatment cycle is 28 days, follow up planned for 1, 3 and 6 months. Overall study period was from January 2007 to November 2012.
Arm/Group | TALL-104 + IM
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TALL-104 + IM (N=3)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TALL-104 + IM (N=3)
Fatigue (General disorders) | 2 (2)
Fever (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema, Limb (Vascular disorders) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal, Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Occular/Visual (Eye disorders) | 1 (1)
Pain, Extremity-Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Headache (Nervous system disorders) | 1 (1)
Pain, Other (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No